CLINICAL TRIAL: NCT04821882
Title: Intravesical Injection of Dextrose to Improve Lower Urinary Tract Symptoms Caused by Chronic Cystitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Juin-Hong Cherng, Assistant Professor, National Defense Medical Center, Taiwan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEXTROSE2019
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Bladder Pain Syndrome; Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Glucose; Long-Term Synaptic Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Healthy participant
- Dextrose treatment (Experimental): IC/PBS patients had been treated by intravesical instillations of hyaluronic acid and/or botox for more than 6 months
  Interventions: Drug: Dextrose

INTERVENTIONS:
Drug: Dextrose — 10% dextrose: 2 mL of 50% dextrose in 10 mL normal saline and injected by 11 sub urothelial injections
  Other Names: Vitagen Inj., Taiwan Biotech Co., Ltd., Taipei, Taiwan
  Arms: Dextrose treatment

SUMMARY:
The pathogenesis of bladder pain syndrome/interstitial cystitis (BPS/IC) is currently unclear. Scholars have put forward different hypotheses, including the function of the extracellular matrix surface of the glycosaminoglycan (GAG) layer, downregulation of tight junction protein, increased urothelial permeability, mast cell activation, neurogenic inflammation, and psychosomatic factors. The symptoms are very similar to severe bladder pain syndrome/interstitial cystitis, and the patients respond to existing medications. In 1956, Dr. George Hackett created a method for treating damaged ligaments and tendons called prolotherapy (proliferation therapy). Prolotherapy is defined as an alternative therapy for musculoskeletal and arthritic pain, including the treatment of irritating substances (such as dextrose, also known as d-glucose) injected into ligaments or tendons to promote the growth of new tissues. There are many clinical trials confirming that proliferation therapy can effectively treat painful musculoskeletal problems. For example, in patients with lateral epicondylitis treated with a solution with a final concentration of 10% dextrose, compared with patients treated with placebo (normal saline), pain and isometric muscle strength improved significantly. A recent literature review also tells that hypertonic glucose proliferation therapy can effectively treat a variety of musculoskeletal diseases.

Hence, this research suggests that dextrose prolotherapy is an affordable and effective pain management strategy in dealing with musculoskeletal neuroinflammation pain in BPS/IC. In order to begin to understand prolotherapy and its therapeutic utility, this study should begin to elucidate the immediate response of prolotherapy in the urology field by investigating the impact of dextrose.

This project is expected to accommodate subjects with BPS/IC, by injecting 10% dextrose into the bladder lining muscles of IC patients and performing various urodynamic tests and questionnaires to evaluate the patient's urinary voiding symptoms and urinary bladder function recovery. Afterward, the expressions of growth factors and cytokines in the urine samples were investigated in an attempt to reveal the mechanism of dextrose prolotherapy in BPS/IC disease.

DETAILED DESCRIPTION:
This project treated 29 male and female subjects (aged over 20 years) with BPS/IC and other chronic inflammation of the bladder. The enrolled subjects were collected from May 2019 to October 2020. The subjects were given intravesical injections of 10% dextrose under intravenous general anesthesia in the operating room: 2 mL of 50% Dextrose (Vitagen Inj., Taiwan Biotech co. ltd., Taipei, Taiwan) was briefly diluted with 10 mL of normal saline and 11 sub urothelial injections (1 mL each site) were performed. The injection needle was inserted into the urothelium at the trigone (1 site), the posterior (6 sites), and the lateral walls (4 sites) of the bladder, using a 23-gauge needle under rigid cystoscopic injection instrument (22-Fr; Knittlingen, Richard Wolf, Germany). No post-injection analgesics were provided to patients. Treatment was repeated based on the patients' condition once every 2 weeks for the first 6 cycles and once every month for the remaining 3 cycles with a maximum of 9 planned therapy cycles up to 6 months. The patients would be followed-up and assessed at each treatment time and up to 1 month after the last treatment. 19 health subjects were also recruited as a healthy control as the comparison.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is aged over 20 years old.
2. The subject was diagnosed as bladder pain syndrome/interstitial cystitis subject with lower urinary tract symptoms, such as frequent urination, urgent urination, bladder pain, etc.

Exclusion Criteria:

1. The subject is aged under 20 years old.
2. Pregnant women.
3. The subject with congenital disorders of the urinary tract.
4. The subject with a urinary tract infection or tumor.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-10-11 (Actual)

PRIMARY OUTCOMES:
Urinary Voiding Symptoms Analysis | 3 days
  Patients were asked to provide a three-day voiding frequency volume chart prior the treatment to record episodes of urinary voiding symptoms including urinary frequency, urgency, and nocturia.
Global Response Assessment (GRA) | Up to 7 months
  GRA examined the overall response to treatment. Patients were requested to rate symptoms on a seven-point centered scale from markedly-, moderately-, and slightly- worse, no change, slightly-, moderately-, and markedly-improved.
International Prostate Symptom Score (IPSS) | Up to 7 months
  The severity of voiding symptoms was evaluated by using the International Prostate Symptom Score (IPSS-TOTAL), and the IPSS-voiding (IPSS-V) and IPSS-storage (IPSS-S) sub-scores were also recorded. There were 7 questions including questions of IPSS-V and IPSS-S.
  The IPSS-V is the sum of the answers to question 1 (incomplete emptying), question 3 (intermittency), question 5 (weak stream), and question 6 (straining to void). Oppositely, the IPSS-S is the sum of the answers to question 2 (frequency), question 4 (urgency), and question 7 (nocturia). The IPSS subscore can be used to evaluate symptom severity or the results of treatment.
  IPSS-TOTAL then took into account the total score from the answers of the questions that can therefore range from 0 to 35 (0-7 mild symptomatic; 8-19 moderately symptomatic; 20-35 severely symptomatic).
Visual Analogue Scale (VAS) | Up to 7 months
  VAS is a pain rating scale which its scores are based on patient self-assessment measures of symptoms that are recorded with a single handwritten mark placed at one point of 10-point along the length of a 10-cm line. The line represents the pain condition, the left end of line scale (0 cm) represents "no pain" and the right end of the scale (10 cm) shows the "worst pain".
O'Leary-Sant Score (OSS) | Up to 7 months
  OSS indexes have eight questions assessing pain and voiding symptoms. OSS is obtained from O'Leary Sant instrument which evaluates a Symptom Index (ICSI with range: 0-20 points) and a Problem Index (ICPI with range: 0-16 points), each of which contains four questions related to urinary and pain symptoms. For each index, the score is calculated by summing the points for each item. A maximal index score of 36 reflects maximal symptom and problem severity.
  The Symptom Index covers various areas, including whether the patient feels the need to urinate with little or no warning, has to urinate more frequently than every 2 hours, needs to get up during the night to urinate, and has pain in the bladder. The Problem Index evaluates other aspects, such as urinary frequency during the day, the urinary frequency at night, the need to urinate with little or no warning, and burning, pain, discomfort, or pressure on the bladder. Both indices evaluate the situation over the previous month.
5-Item Brief Symptom Rating Scale (BSRS-5) | Up to 7 months
  BSRS-5 evaluated the quality of life of patients. It contained five items of a self-administered questionnaire that is derived from the 50-item brief symptom rating scale. The score for each item ranges from 0 to 4 (from not at all to extremely). A total score on the BSRS-5 above 14, between 10 and 14, and between 6 and 9 indicated severe, moderate, and mild symptoms, respectively.
5-item Female Sexual Function Index (FSFI-5) | Up to 7 months
  FSFI-5 was performed to assess the sexual dysfunction possibility of female patients. FSFI-5 contained item-by-item combinations of the 5 domains of sexual "desire", "arousal", "lubrication", "orgasm", and "satisfaction". The 5 items were derived from 19 items of FSFI questionnaire.
Luminex Assay of Growth Factors | Up to 7 months
  Urine samples were collected and stored at 4°C until analysis. Samples were analyzed for the presences of 4 analytes: epidermal growth factor (EGF), hepatocyte growth factor (HGF), placental growth factor-1 (PIGF-1), and vascular endothelial growth factor-D (VEGF-D). Their concentration was measured using a Growth Factor 11-Plex Human ProcartaPlex™ Panel assay kit with magnetic beads (EPX110-12170-901, Thermo Fisher Scientific, MA, USA) and examined with an automated immunoassay analyzer (Luminex™ 100 IS System, Luminex, TX, USA) and the accompanying ProcartaPlex Analyst Software 1.0 (Thermo Fisher Scientific, MA, USA) according to the manufacturer's instructions.
Luminex Assay of Cytokine Assay | Up to 7 months
  The levels of serum cytokines [interleukin-6 (IL-6), IL-10, IL-12p70, IL-13, IL-17F, and IL-27] in blood samples were detected using a magnetic bead-based multiplex immunoassay MILLIPLEX MAP Human Th17 Magnetic Bead Panel (Merck KGaA, Darmstadt, Germany) according to the manufacturer's protocol. The MAGPIX® System reader was used to acquire the data of cytokines, which was output as concentration (pg/mL) using the Belysa™ Immunoassay Curve Fitting Software (Merck KGaA, Darmstadt, Germany).
Statistics Analysis | Up to 7 months
  Urinary voiding symptoms analysis, the score of questionnaires (GRA, IPSS-TOTAL, IPSS-V, IPSS-S, VAS, ICSI, ICPI, BSRS5, and FSFI5), Luminex assay result of growth factors and cytokines assay were compared between and after treatment. Results are presented as mean values plus or minus standard deviations. Statistical comparisons between the groups were tested using a chi-square test for categorical variables, and an independent t test or a Wilcoxon test for nonparametric data was used for multiple comparisons. The correlation analysis and coefficient statistical method were performed for comparing VAS questionnaire and growth factor relation. A P value of <0.05 was considered statistically significant. Statistical analyses were performed using SPSS 18.0 statistical software (SPSS Inc., IL, USA).

CONTACTS AND LOCATIONS:
Locations (1):
- National Defense of Medical Center, Tri-Service General Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Meng E, Hsu YC, Chuang YC. Advances in intravesical therapy for bladder pain syndrome (BPS)/interstitial cystitis (IC). Low Urin Tract Symptoms. 2018 Jan;10(1):3-11. doi: 10.1111/luts.12214. PMID 29341502
- [Background] Hanno PM. Campbell-Walsh Urology. In: Wein AJ, Kavoussi LR, Partin AW, Peters C, editors. Bladder pain syndrome (interstitial cystitis) and related disorder. 1. Eleventh edition. ed. Philadelphia. PA: Elsevier. 2016; p. 334-70.
- [Background] Middela S, Pearce I. Ketamine-induced vesicopathy: a literature review. Int J Clin Pract. 2011 Jan;65(1):27-30. doi: 10.1111/j.1742-1241.2010.02502.x. PMID 21155941
- [Background] Tsai TH, Cha TL, Lin CM, Tsao CW, Tang SH, Chuang FP, Wu ST, Sun GH, Yu DS, Chang SY. Ketamine-associated bladder dysfunction. Int J Urol. 2009 Oct;16(10):826-9. doi: 10.1111/j.1442-2042.2009.02361.x. Epub 2009 Jul 29. PMID 19659678
- [Background] Chu PS, Ma WK, Wong SC, Chu RW, Cheng CH, Wong S, Tse JM, Lau FL, Yiu MK, Man CW. The destruction of the lower urinary tract by ketamine abuse: a new syndrome? BJU Int. 2008 Dec;102(11):1616-22. doi: 10.1111/j.1464-410X.2008.07920.x. Epub 2008 Aug 1. PMID 18680495
- [Background] Shahani R, Streutker C, Dickson B, Stewart RJ. Ketamine-associated ulcerative cystitis: a new clinical entity. Urology. 2007 May;69(5):810-2. doi: 10.1016/j.urology.2007.01.038. PMID 17482909
- [Background] Hackett GS, Hemwall G, Montgomery GJS, IL, Charles C. Thomas. Ligament and Tendon Relaxation. 1956.
- [Background] Scarpone M, Rabago DP, Zgierska A, Arbogast G, Snell E. The efficacy of prolotherapy for lateral epicondylosis: a pilot study. Clin J Sport Med. 2008 May;18(3):248-54. doi: 10.1097/JSM.0b013e318170fc87. PMID 18469566
- [Background] Seven MM, Ersen O, Akpancar S, Ozkan H, Turkkan S, Yildiz Y, Koca K. Effectiveness of prolotherapy in the treatment of chronic rotator cuff lesions. Orthop Traumatol Surg Res. 2017 May;103(3):427-433. doi: 10.1016/j.otsr.2017.01.003. Epub 2017 Feb 16. PMID 28215611
- [Background] Sit RW, Chung VCh, Reeves KD, Rabago D, Chan KK, Chan DC, Wu X, Ho RS, Wong SY. Hypertonic dextrose injections (prolotherapy) in the treatment of symptomatic knee osteoarthritis: A systematic review and meta-analysis. Sci Rep. 2016 May 5;6:25247. doi: 10.1038/srep25247. PMID 27146849
- [Background] Hauser RA, Lackner JB, Steilen-Matias D, Harris DK. A Systematic Review of Dextrose Prolotherapy for Chronic Musculoskeletal Pain. Clin Med Insights Arthritis Musculoskelet Disord. 2016 Jul 7;9:139-59. doi: 10.4137/CMAMD.S39160. eCollection 2016. PMID 27429562